CLINICAL TRIAL: NCT00610493
Title: A Phase I Trial of Bevacizumab and Temsirolimus in Patients With Advanced Malignancy
Brief Title: Bevacizumab and Temsirolimus in Patients With Advanced Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0668; NCI-2012-01750 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Bevacizumab; Temsirolimus; Avastin; Torisel; CCI-779; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; dynamic contrast-enhanced magnetic resonance imaging; DCE; magnetic resonance imaging; MRI
MeSH Terms: interventions — Bevacizumab; temsirolimus; Biopsy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bevacizumab + Temsirolimus (Experimental): Bevacizumab 5 mg/kg By Vein Over 90 Minutes on Day 1 of Each 21 Day Cycle. Temsirolimus 5 mg By Vein Over 30-60 Minutes on Days 1, 8, 15 of Each 21 Day Cycle. First tumor biopsy during screening visit and Second at the end of Cycle 1. DCE-MRI (dynamic contrast-enhanced magnetic resonance imaging) scan during screening visit, at 24-48 hours after the start of Cycle 1, and at the end of Cycle 1.
  Interventions: Drug: Bevacizumab; Drug: Temsirolimus; Procedure: Additional Blood Drawn; Procedure: Biopsy; Procedure: DCE-MRI Scan

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg By Vein Over 90 Minutes on Day 1 of Each 21 Day Cycle
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Temsirolimus — 5 mg By Vein Over 30-60 Minutes on Days 1, 8, 15 of Each 21 Day Cycle
  Other Names: Torisel; CCI-779
Procedure: Additional Blood Drawn — 2 teaspoons each time: 4xDay Cycle 1 after start of first infusion; at Day 8 of Cycle 1; at Day 15 of Cycle 1; and at end of Cycle 1.
Procedure: Biopsy — First tumor biopsy during screening visit and Second at the end of Cycle 1
Procedure: DCE-MRI Scan — DCE-MRI (dynamic contrast-enhanced magnetic resonance imaging) scan during screening visit, at 24-48 hours after the start of Cycle 1, and at the end of Cycle 1
  Other Names: imaging scans; dynamic contrast-enhanced magnetic resonance imaging; DCE; magnetic resonance imaging; MRI

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Avastin (bevacizumab) and Torisel (temsirolimus) that can be given, in combination, to patients with advanced cancer that has spread or is unable to be surgically removed. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels that supply nutrients necessary for tumor growth.

Temsirolimus is designed to block the growth of cancer cells, which may cause cancer cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of bevacizumab and temsirolimus combined, based on when you joined this study. Up to 13 dose levels of the study drug combination will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug combination is found.

If you choose to enroll in the expansion group of patients being treated at the highest tolerable dose of the study drug combination found, you will be required to undergo added testing, as follows:

* You will have additional blood drawn (about 2 teaspoons each time) during Cycle 1. This blood will be drawn before you begin taking the study drugs; on Day 1 at about 1, 4, 8, and 24 hours after the start of your first infusion; at Day 8 of Cycle 1; at Day 15 of Cycle 1; and at the end of Cycle 1. The blood will be used to see how the study drug combination acts in the body and to learn its effect on cancer cells.
* You will have 2 tumor biopsies performed. These samples will be used to see how the study drug combination acts in the body and to learn its effect on cancer cells. These tumor biopsies will be performed during the screening visit and at the end of Cycle 1. To perform a tumor biopsy, the affected area is numbed with anesthetic and some or all of the tumor tissue is removed with a small knife.
* You will have extra imaging scans performed and used to see how the study drug combination may be affecting blood vessels that supply nutrients and oxygen to cancer. A DCE-MRI scan will be performed during the screening visit, at 24-48 hours after the start of Cycle 1, and at the end of Cycle 1. Like a regular MRI scan, the DCE-MRI scan involves passing part or all of the body into a long, narrow tube scanner that is open at both ends.

Study Drug Administration:

Bevacizumab and temsirolimus will be given in "cycles." Cycles will be about 21 days long or longer, depending on any side effects you may experience.

Bevacizumab is given by vein on Day 1 of each cycle. On Day 1 of Cycle 1, you will receive it over 90 minutes. If you tolerate it well in Cycle 1, you will receive it over 60 minutes in Cycle 2. If you tolerate it well in Cycle 2, you will receive it over 30 minutes in Cycle 3. It will continue to be given over 30 minutes in Cycle 4 and further cycles, as long as you still tolerate it well. Also, if the first dose is well tolerated, you may be given the remaining doses of Bevacizumab in the doctor's office in or near your hometown.

Temsirolimus is given by vein on Days 1, 8, and 15 of each cycle. During Day 1 of Cycle 1, you will receive it over 60 minutes. If you tolerate it well on Day 1 of Cycle 1, it will be given over 30 minutes on Days 8 and 15 of Cycle 1 and over 30 minutes in further cycles, as long you still tolerate it well. Also, if the first dose is well tolerated, you may be given the remaining doses of Temsirolimus in the doctor's office in or near your hometown.

Study Visits:

You will have a physical exam and blood drawn (about 1 tablespoon each time) for routine tests once between Days 7 and 14 during Cycle 1. During the rest of the cycles, you will have a physical exam and blood drawn (about 1 tablespoon each time) for routine tests once every 3 weeks. The status of the disease will be checked by a CT or MRI scan after every 2 cycles, starting after Cycle 2.

Length of Study Participation:

You may continue to receive additional cycles of the study drugs, unless the cancer gets worse or intolerable side effects occur. In that case, you will be taken off study.

Once your participation is over in this study, you will receive standard-of-care follow-up for the disease.

This is an investigational study. Bevacizumab and temsirolimus are commercially available. Bevacizumab is FDA approved for the treatment of colorectal cancer and a type of lung cancer. Temsirolimus is FDA approved for the treatment of kidney cancer that has spread. The combination of bevacizumab and temsirolimus is not FDA approved. At this time, it is being used in research only.

Up to 183 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that induces a CR rate of at least 10% or improves survival by at least three months.
2. Patients should be at least four weeks from the last day of therapeutic radiation or cytotoxic chemotherapy or from antibody therapy, or at least five half-lives from non-cytotoxic targeted or biologic therapy. Patients may have received palliative radiation immediately before (or during) treatment provided radiation is not to the only target lesion available.
3. ECOG performance status </= 2 (Karnofsky >/= 60%).
4. Patients must have allowable organ and marrow function defined as: absolute neutrophil count >/= 1,000/mL; platelets >/=50,000/mL; creatinine </= 3 X ULN; total bilirubin </= 3.0; AST(SGOT)/ALT(SGPT) </= 5 X ULN; fasting level of total cholesterol of no more than 350mg/dL; triglyceride level of no more than 400mg/dL.
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose.
6. Ability to understand and the willingness to sign a written informed consent document
7. Patients may not be receiving any other investigational agents and/or any other concurrent anticancer agents or therapies.

Exclusion Criteria:

1. Patients with hemoptysis within 28 days prior to entering the study.
2. Patients with clinically significant unexplained bleeding within 28 days prior to entering the study
3. Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg on medication).
4. Patients with clinically significant cardiovascular disease: - History of CVA within 6 months - Myocardial infarction or unstable angina within 6 months - Unstable angina pectoris
5. Pregnant or lactating women.
6. History of hypersensitivity to bevacizumab, murine products, or any component of the formulation.
7. History of hypersensitivity to Temsirolimus or its metabolites (including sirolimus), polysorbate 80, or to any component of the formulation
8. Patients that are taking CYP3A4 inducers and/or inhibitors. Please see section 3.2 in the protocol for details. If a patient has a history of taking CYP3A4 inducers and/or inhibitors prior to enrollment on the protocol, it is strongly recommended that the patient stops the drug and waits at least 5 half-lives of said drug before initiating therapy on protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2008-01-25 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days
  Maximum tolerated dose defined as the dose level below the dose at which two of six patients experience drug-related dose limiting toxicity in the first cycle.

SECONDARY OUTCOMES:
Anti-Tumor Efficacy | Baseline, 24-48 hours after the start of Cycle 1, and at the end of Cycle 1. Cycles are 21 days.
  Anti-tumor efficacy of each combination determined by objective response per RECIST and WHO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Piha-Paul, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org